CLINICAL TRIAL: NCT02975024
Title: Blood Flow Analysis of the Human Mucosa After Vestibuloplasty Procedures
Status: Completed | Type: Observational
Sponsor: Semmelweis University (Other)
Collaborators: Hungarian Scientific Research Fund (Unknown)
Responsible Party: Principal Investigator, Dr. Vag Janos, associate professor, Semmelweis University
Other Study IDs: 3/2013
Record Dates: First submitted 2016-11-16; First posted 2016-11-29 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Mucogingival Defect
Keywords: mandibular vestibuloplasty; wound healing; microcirculation; Laser Speckle Contrast Imager; Mucograft; strip gingival graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mucograft: Laser speckle contrast imaging of the oral mucosa and wound fluid measurement and quantitative determination of VEGF after mandibular vestibuloplasty. Individuals of this pre-defined group are candidates of vestibuloplasty, where the keratinized gingiva will be enlarged by a combination of apically repositioned split thickness flap with a xenogeneic collagen matrix (Mucograft).
  Interventions: Device: laser speckle contrast imaging of the oral mucosa; Device: wound fluid measurement; Device: quantitative determination of VEGF
- strip gingival graft + Mucograft: Laser speckle contrast imaging of the oral mucosa and wound fluid measurement and quantitative determination of VEGF after mandibular vestibuloplasty. Individuals of this pre-defined group are candidates of vestibuloplasty, where the keratinized gingiva will be enlarged by a combination of apically repositioned split thickness flap with a strip gingival graft and a xenogeneic collagen matrix (Mucograft). The strip gingival graft is harvested from the patient's palate.
  Interventions: Device: laser speckle contrast imaging of the oral mucosa; Device: wound fluid measurement; Device: quantitative determination of VEGF

INTERVENTIONS:
Device: laser speckle contrast imaging of the oral mucosa — Non-invasive method to measure tissue blood perfusion applied for oral mucosa
  Other Names: LSCI Perimed PSI
Device: wound fluid measurement — Wound fluid at the wound margin is collected using filter strip and volumetrically measured by Periotron 8010 instrument.
  Other Names: Periotron 8010
Device: quantitative determination of VEGF — For the quantitative determination of VEGF in the fourth day wound fluid sample the Human VEGF Quantikine ELISA Kit will be used.
  Other Names: Human VEGF Quantikine ELISA Kit

SUMMARY:
Apply the LSCI for follow-up the postoperative microcirculation after surgical procedures to enlarge keratinized gingiva in order to characterize the kinetics of the blood flow changes during wound healing in human subjects.

DETAILED DESCRIPTION:
Vestibuloplasty is the common name of those procedures designed to widen the zone of attached gingiva. The apically repositioned split thickness flap with a xenogeneic collagen matrix or with a combination of strip gingival graft and a xenogeneic collagen matrix are frequently used surgical techniques, however no data are available, how these graft tissues affect the microcirculation of the healing gingiva.

LSCI is a non-invasive, two dimensional method to evaluate microcirculation of different tissues. This new method let us monitor the entire surgical area real-time during the healing period.

The aim of the present study is to define blood flow patterns, which might characterize the wound healing of such surgical procedures during the first 6 months of healing in order to facilitate treatment.

ELIGIBILITY:
Ages Eligible for Study: 18 Years to 45 Years Genders Eligible for Study: Both Accepts Healthy Volunteers: Yes

Inclusion Criteria:

• clinical diagnosis of inadequate width of keratinized gingiva at the mandibular front region

Exclusion Criteria:

* pregnancy
* heavy smoking
* general diseases
* taking medications or having treatments which have an effect on mucosal healing in general (e.g. steroids, anti-inflammatory drugs)
* taking any other medications in the last three months (except contraceptives)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Caucasians subjects presenting multiple Miller Class I. and II. gingival recessions (Multiple Adjacent Recession Type Defects, MARTD) were recruited in the Department of Periodontology in Semmelweis University.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Postoperative blood flow changes of the oral mucosa | 6 months after surgery
  Blood flow changes are measured by Laser Speckle Contrast Imager (LSCI) after mandibular vestibuloplasty. The scale is an arbitrary unit (0-3000 LSPU) and the relative changes to the surgically unaffected surrounding mucosa measurements are calculated. Postoperative follow-up time-points are: 1, 2, 3, 4, 5, 6, 7, 9, 11, 14, 21, 28 days, and 2, 3, 4, 5, 6 months. The apically repositioned split thickness flap is combined either with a Mucograft alone, or with a combination of autologous strip gingival graft and Mucograft. The differences in postoperative blood flow changes are compared between the two surgical techniques.

SECONDARY OUTCOMES:
Wound fluid volume measurement | 14 days after surgery
  Wound fluid sample is collected using a filter strip to withdraw the fluid around the wound. The filter strip is then inserted into Periotron 8010 instrument to score the volume on the paper. Scores are measured in an arbitrary unit. Postoperative follow-up time-points are: 1, 2, 3, 4, 5, 6, 7, 9, 11, 14 days. The apically repositioned split thickness flap is combined either with a Mucograft alone, or with a combination of autologous strip gingival graft and Mucograft. The differences in postoperative wound fluid changes are compared between the two surgical techniques.
Evaluation of the periodontal parameters at teeth at the surgical site: a composite outcome measure consisting of multiple measures. | Pre- and six month postoperative
  Periodontal parameters are evaluated using a periodontal probe and will be expressed in mm. The following will be assessed at each tooth at the surgical site: probing depth, depth and width of recession, papilla height, and width and thickness of the keratinized gingiva. Surgical area is also measured apico-coronally and mesio-distally, during the whole follow-up period.
Quantitative determination of Vascular Endothelial Growth Factor (VEGF) of the wound fluid | 4 days after surgery
  Wound fluid sample for VEGF is collected at the fourth postoperative day. For the quantitative determination of VEGF in samples the Human VEGF Quantikine ELISA Kit will be used. The apically repositioned split thickness flap is combined either with a Mucograft alone, or with a combination of autologous strip gingival graft and Mucograft. The differences in postoperative wound fluid level of VEGF (expressed in conc pg/mL) are compared between the two surgical techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Janos Vag, Principal Investigator — Semmelweis University, Dept. of Conservative Dentistry
Locations (1):
- Janos Vag, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No